CLINICAL TRIAL: NCT03184506
Title: Effect of Pre-warming on Perioperative Hypothermia and Shivering During Holmium Laser Enucleation of the Prostate (HoLEP) Under Spinal Anesthesia
Brief Title: Effect of Pre-warming on Perioperative Hypothermia During HoLEPunder Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Jun joohyun, assistant professor, Hallym University Kangnam Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017-05-002
Record Dates: First submitted 2017-06-05; First posted 2017-06-12 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2017-06

CONDITIONS: Hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Sham Comparator)
  Interventions: Other: no warming
- pre-warming group (Active Comparator)
  Interventions: Other: pre-warming

INTERVENTIONS:
Other: pre-warming — On arrival at the preoperative care unit, assignments were determined using an opaque sealed envelope opened by investigator with no clinical involvement in the study. In the pre-warming group, the forced-air blanket (COVIDIEN™ WarmTouch™ Full Body/Multi Access Blanket, Covidien Ilc, Mansfield, MA, USA) was positioned over the whole body except head and neck, covered by cotton blanket. Forced air warmer (COVIDIEN™ WarmTouch™ WT6000 Warming Unit, Covidien Ilc, Mansfield, MA, USA) was set to 'high level' (45℃) during 20 min. During the warming procedure, patients were asked every 5 min about their thermal comfort; if they felt overheated, the warmer was lowered to 41℃
  Arms: pre-warming group
Other: no warming — patients were covered only with two layers of cotton blanket
  Arms: control group

SUMMARY:
Inadvertent perioperative hypothermia is an unintentional drop in core body temperature below 36°C. Intraoperative hypothermia can lead to serious clinical complications such as, myocardial ischemia, coagulopathy, immunosuppression, and surgical wound infection. Hypothermia develops easily during surgeries that require irrigation fluid, such as laparoscopic surgery and transurethral resection of the prostate. Although isothermic irrigation fluid was suggested to prevent perioperative hypothermia, it can be difficult to warm a large volume of irrigation fluid.

Re-distribution after induction of anesthesia is the most important cause of perioperative hypothermia. The extent of re-distribution is proportional to the gradient between the core and peripheral compartments. Pre-warming increases the heat content of the peripheral thermal compartment, reducing the gradient for redistribution. Recently, A recent-meta analysis suggested that as a single strategy, preoperative forced air warming had significant benefits than other warming methods. Also, it was reported that only 20 (or even 10) min of pre-warming mostly prevented patients from perioperative hypothermia under general anesthesia. However, few studies have examined whether short time pre-warming can reduce hypothermia due to a large amount of irrigation fluid during surgery under spinal anesthesia.

The purpose of this study is to assess whether the application of preoperative forced air warming set to high temperature (> 43°C) for brief period can prevent hypothermia or shivering during procedures requiring large volumes of cold irrigation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with ASA physical status I-III, aged 50 - 80 years, undergoing HoLEP under spinal anesthesia

Exclusion Criteria:

* preoperative body temperature of more than 37.2°C preexisting severe cardiovascular, respiratory and endocrinal disease on anticoagulant therapy

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
core temperature | on admission to PACU
  taken in the same ear using an infrared tympanic thermometer (ThermoScan IRT 1020; Braun, Germany), and the highest reading from three consecutive measurements was recorded.

SECONDARY OUTCOMES:
the incidence of perioperative hypothermia | at baseline (preoperative care unit), on arrival at the OR, every 10 minutes after spinal anesthesia, and on admission to PACU 1 hour
  Hypothermia defined as a core temperature less than 36.0°C in according to the current guideline. The number of patients who became hypothermic at each time was recorded.
the incidence of shivering | on arrival at the OR, at every 30 minutes after spinal anesthesia, on admission to PACU, and then every 30 minutes for 1 hour.
  graded using 4 point scale (0 = no shivering; 1 = shivering localized to the core and neck; 2 = shivering including the upper extremities; and 3 = total body shivering)
Thermal comfort | on arrival at the OR, at every 30 minutes after spinal anesthesia, on admission to PACU, and then every 30 minutes for 1 hour.
  evaluated using a numeric rating scale: 0 was defined as 'extremely cold', 5 as 'thermally neutral', and 10 as 'extremely hot'
core temperature | at baseline (preoperative care unit), on arrival at the operation room, every 30 minutes after spinal anesthesia
  taken in the same ear using an infrared tympanic thermometer (ThermoScan IRT 1020; Braun, Germany), and the highest reading from three consecutive measurements was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Kangnam Sared heart Hospital, Seoul, Yeongdeungpo-gu, South Korea

REFERENCES:
- [Derived] Jun JH, Chung MH, Kim EM, Jun IJ, Kim JH, Hyeon JS, Lee MH, Lee HS, Choi EM. Effect of pre-warming on perioperative hypothermia during holmium laser enucleation of the prostate under spinal anesthesia: a prospective randomized controlled trial. BMC Anesthesiol. 2018 Dec 22;18(1):201. doi: 10.1186/s12871-018-0668-4. PMID 30579334